CLINICAL TRIAL: NCT05561790
Title: Determination of Optimal Sleep Treatment Elements (The DOSE Project)
Brief Title: Determination of Optimal Sleep Treatment Elements - Pilot
Acronym: DOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry); Enversion A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-051-000001-2099-1
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-09

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Administration of sleep hygiene, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy.
  Interventions: Behavioral: eCBT-I
- Control (No Intervention): Waitlist control (sleep diary only); access to treatment after final measurement

INTERVENTIONS:
Behavioral: eCBT-I — Automated digital administration of sleep hygiene, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy modules via mobile or web application, lasting approximately six weeks.
  Arms: Intervention

SUMMARY:
Previous research has shown the efficacy of (combinations of) individual components of cognitive behavioral therapy for insomnia (CBT-I), namely sleep hygiene education, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy. However, their relative effects, i.e., their effects in direct comparison with each other, are yet to be assessed.

In this pilot study, a smartphone and web application developed to treat insomnia using these treatment components will be tested.

Two future studies will investigate the components' relative efficacy in order to identify the most effective component or combination of components for digitized treatment of chronic insomnia by means of the Multiphase Optimization Strategy (MOST), and verify this intervention's effect in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
As a pilot study for a Multiphase Optimization Strategy (MOST) study, the current study will assess the effects of a newly developed smartphone and web application for digitized cognitive behavioural therapy for insomnia (eCBT-I). All treatment components, i.e., sleep hygiene education, sleep optimization, stimulus control therapy, deactivation/relaxation training, and cognitive therapy, will be tested in order to receive feedback on the functioning of the application as well as to get an initial impression of possible treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Individuals who report moderate-to-severe insomnia symptoms (a score ≥10 on the Insomnia Severity Index, ISI)
* Individuals with access to a smartphone or computer with internet connection
* Individuals who report sufficient technological proficiency (e.g., ability to download apps)

Exclusion Criteria:

* Children (<18 years)
* Individuals who report mild or no clinically relevant insomnia symptoms (a score <10 on the ISI)
* Individuals who have a shift-work schedule or are on maternity/paternity leave, if this impacts their sleep quality or amount of sleep
* Individuals who are unable to read Danish
* Individuals who report severe physical or psychological comorbidity with known effects on sleep (e.g., psychosis, cardiovascular disease, cancer, COPD)
* Individuals who report other diagnosed sleep or circadian rhythm disorders (e.g., sleep apnea, narcolepsy)
* Individuals who have previously used the "Hvil®"-app, e.g., during the beta test phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Insomnia severity post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Insomnia Severity Index (ISI), with scores ranging from 0 to 28, where higher scores indicate higher insomnia severity, and a score equal to or above 10 indicates clinical significance.

SECONDARY OUTCOMES:
Sleep diary assessed sleep efficiency (SE) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Based on the Consensus Sleep Diary (CSD) which measures bedtime, rise-time, sleep- and waking time, sleep onset latency, wakefulness after initial sleep onset, allowing for total sleep time, total time in bed, and sleep efficiency to be calculated. SE is calculated as the proportion of time spent asleep out of time spent in bed in percent (TST/TiB*100).
Sleep diary assessed sleep onset latency (SOL) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Assessed with the Consensus Sleep Diary (CSD)
Sleep diary assessed wake after sleep onset (WASO) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Assessed with the Consensus Sleep Diary (CSD)
Sleep diary assessed nocturnal awakenings (NA) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Assessed with the Consensus Sleep Diary (CSD)
Sleep diary assessed total sleep time (TST) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Based on the Consensus Sleep Diary (CSD) which measures bedtime, rise-time, sleep- and waking time, sleep onset latency, wakefulness after initial sleep onset, allowing for total sleep time to be calculated.
Sleep diary assessed time in bed (TiB) at end of intervention | Approximately 10 weeks after study entry (randomization)
  Based on the Consensus Sleep Diary (CSD) which measures bedtime, rise-time, sleep- and waking time, sleep onset latency, wakefulness after initial sleep onset, allowing for time in bed to be calculated.
Daytime fatigue post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-Fatigue), which covers physical fatigue, functional fatigue, and social consequences of fatigue.
Cognitions about sleep post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16).
Psychological distress post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Depression, Anxiety, and Stress Scales-21 (DASS-21), which evaluates the constructs depression, anxiety, and stress on sub-scales.
Usability post-intervention | 11 weeks after study entry (randomization)
  Assessed with the mHealth App Usability Questionnaire (MAUQ).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, DMSc, MSc, Principal Investigator — Aarhus University, Aarhus University Hospital
Locations (1):
- Aarhus University, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the study will be made available in an irreversibly anonymized form. However, only data of those participants can be shared who have explicitly given consent to this as part of their informed consent to study participation. This means that it may not be possible to share all data underlying a certain publication.
  Data will be shared exclusively for research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No later than six months after publication, no end date.
Access Criteria: Data will be shared exclusively with other researchers and for research purposes only. Researchers requesting the data will have to provide a methodologically sound research proposal clarifying how the data will be used and for what purpose.